CLINICAL TRIAL: NCT02615483
Title: Lumbar Spinal Fusion - Web-based Platform Targeting Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Janni Stroem, Ph.D. - Student, Central Jutland Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 654902
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Lumbar Spine Fusion; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web-based platform (Experimental): Access to a web-based platform
  Interventions: Other: Web-based platform
- Control (No Intervention): Conventional

INTERVENTIONS:
Other: Web-based platform — The WP is based on a conducted literature review and results form a previous study conducted in the regional context of the study. Information on the WP is animated based on the current literature stating that educative animation video optimises patients' acquisition of knowledge. The intention is to offer the patients the advantages in gaining knowledge in familiar surroundings and at a pace matching their needs and wishes.
  The WP contains animated and written information mirroring the course of treatment, frequently asked questions and answers, it contains animated training support, a diary in order to keep track of training and development of pain and finally a social feature, a web-café.
  Arms: Web-based platform

SUMMARY:
The purpose of the present study is to investigate the effect of a Web- based Platform (WP) on anxiety and depression and health economics among patients undergoing lumbar spine fusion (LSF).

DETAILED DESCRIPTION:
This study will seek to reduce pre- and postoperative anxiety, depression and functional impairments using alternative cognitive and educative methods, targeting the underlying factors for development of anxiety and depression.

It is known that there is a rationale behind using Cognitive Behavioural Therapy (CBT) in order to reduce pre- and postoperatively anxiety and depression. The main assumption within CBT is that patients´ perceptions create their thoughts and beliefs, which influence their feelings and subsequently their behaviour. The features of WP in this study will seek in several ways to exceed this expected behaviour modification. The preliminary choices of features on the WP are made in order to prevent catastrophic images and thereby reduce anxiety and depression. The WP will offer patients non-catastrophic images through animated information mirroring the course of treatment, which will aim to influence their beliefs, feelings and their behaviour.

To examine the effect of the WP versus conventional information and course of rehabilitation, on patients' degree of anxiety and depression, a randomized controlled trial will be preformed. A total of 114 patients scheduled for elective instrumented LSF will be included and randomly assigned to the control group or to the intervention group receiving access to the WP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to have a one-three level instrumented Lumbar Spinal Fusion

Exclusion Criteria:

* Age below 18, known psychiatric disorder, prior LSF, as the success rates of re-operations are found as low as 35%, inability to communicate in Danish and finally patients with no internet connection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-11; Primary Completion 2018-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depression | 3 months after surgery
  The change in anxiety and depression measures by Hospital Anxiety and Depression Scale (HADS)

SECONDARY OUTCOMES:
Functional outcome | 3, 6,12 months after surgery
  Oswestry Disability Index (ODI)
Self-perceived health status | 3, 6, 12 months after surgery
  EQ-5D
Back and leg pain | 3, 6, 12 months after surgery
  Low Back Pain Rating Scale (LBPRS)
Anxiety and Depression | 6, 12 months after surgery
  HADS

CONTACTS AND LOCATIONS:
Overall Officials: Claus V. Nielsen, professor, Principal Investigator — Institute of Publich health, Aarhus University
Locations (1):
- Centre og Elective Surgery, Regional Hospital Silkeborg, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data